CLINICAL TRIAL: NCT01130909
Title: A Phase I, Randomized, Double-Blind, Four-way Cross-over Study in Healthy Subjects to Assess Quantitative Electroencephalography (qEEG) Parameters After the Administration of Ketamine, Two Doses of AZD6765 and Placebo
Brief Title: A Blinded, Four-Way Crossover in Healthy Subjects to Assess EEG After Administration of Ketamine, Placebo and AZD6765
Acronym: AZD6765 EEG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The benefit of halting the study to analyze the available data outweighs the benefit of delaying the analysis to include data from remaining treatment periods
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D2285M00008
Record Dates: First submitted 2010-05-19; First posted 2010-05-26 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Healthy; Effect of a single dose on gamma-band qEEG
MeSH Terms: interventions — AZD6765; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD6765 75 mg (Experimental)
  Interventions: Drug: AZD6765
- AZD6765 150 mg (Experimental)
  Interventions: Drug: AZD6765
- Ketamine 0.5 mg/kg (Active Comparator)
  Interventions: Drug: Ketamine
- 125 mL sterile NaCl 0.9% (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6765 — 75 mg
  Arms: AZD6765 75 mg
Drug: AZD6765 — 150 mg
  Arms: AZD6765 150 mg
Drug: Ketamine — 0.5 mg/kg
  Arms: Ketamine 0.5 mg/kg
Drug: Placebo — 125 mL sterile NaCl 0.9%
  Arms: 125 mL sterile NaCl 0.9%

SUMMARY:
This study will provide data to support preclinical to clinical translation by aligning preclinical and clinical efficacy assay with dose dependent changes in EEG.

DETAILED DESCRIPTION:
A Phase I, Randomized, Double-Blind, Four-way Cross-over Study in Healthy Subjects to Assess Quantitative Electroencephalography (qEEG) parameters after the administration of ketamine, two doses of AZD6765 and Placebo

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30 Non-smoker for at least 4 weeks

Exclusion Criteria:

* Any clinically relevant acute or chronic disease
* History of substance abuse Hypersensitivity to ketamine

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
qEEG assessed through the gamma bands | Day 1 of each treatment period at Predose, 0.25h, 1h, 1.25h, 3h and 8h

SECONDARY OUTCOMES:
Pupil Size - to assess the relationship between qEEG and pupil size | Day 1 of each treatment period at Predose, 0.25h, 1h, 1.25h, 3h, and 8h
Electronystagmography - to assess the relationship between qEEG and spontaneous nystagmus. | Day 1 of each treatment period at Predose, 1h, 3h, and 8h
Bond/Lader scales and eVAS - to assess the subject's alertness, calmness and contentment | Day 1 of each treatment period at Predose, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, and 8h

CONTACTS AND LOCATIONS:
Overall Officials: Albena Patroneva, MD, Study Director — AstraZeneca; Francine Santoro, Principal Investigator — Forenap
Locations (1):
- Research Site, Rouffach, France

REFERENCES:
- [Derived] Sanacora G, Smith MA, Pathak S, Su HL, Boeijinga PH, McCarthy DJ, Quirk MC. Lanicemine: a low-trapping NMDA channel blocker produces sustained antidepressant efficacy with minimal psychotomimetic adverse effects. Mol Psychiatry. 2014 Sep;19(9):978-85. doi: 10.1038/mp.2013.130. Epub 2013 Oct 15. PMID 24126931
- See also: D2285M00008 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1245&filename=D2285M00008_Clinical_Study_Report_Synopsis.pdf